CLINICAL TRIAL: NCT02811133
Title: Inositol for Comorbid Anxiety in Children and Adolescents With Bipolar Disorder
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding terminated
Sponsor: Ronald M. Glick, MD (Other)
Collaborators: The Fine Foundation (Unknown); Jarrow Formulas Inc (Industry)
Responsible Party: Sponsor-Investigator, Ronald M. Glick, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100221
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Bipolar Disorder; Anxiety Disorders; Anxiety
Keywords: inositol
MeSH Terms: conditions — Bipolar Disorder; Anxiety Disorders | interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inositol (Experimental): Subjects will receive inositol
  Interventions: Drug: Inositol

INTERVENTIONS:
Drug: Inositol — Subjects will receive inositol
  Other Names: Myoinositol

SUMMARY:
This is an open trial that seeks to determine the safety and tolerability of using inositol for children and adolescents with bipolar disorder and comorbid anxiety disorders with an exploration of efficacy and dose-response.

DETAILED DESCRIPTION:
Anxiety disorders are common comorbidities among children and adolescents with bipolar disorder. Treatment with standard pharmacologic agents may worsen mood problems or lead to drug dependency. Inositol has shown benefits for bipolar depression in adults. This is an open multi-case control study. The investigators will enroll 20 children and adolescents ages 8-17 treated at the Child and Adolescent Bipolar Services (CABS) at Western Psychiatric Institute and Clinic. Participants' involvement will be 14 weeks, including the initial titration of the supplement, maintenance, and taper. Primary outcomes will include standard measures of mood and anxiety. Also, physiologic measures including body mass index and bedside glucose will be followed.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence in the medical record confirming the DSM-V diagnosis of bipolar disorder. If this documentation is not in the record, then the appropriate sections of K-SADS will be administered to confirm the diagnosis.
2. Evidence in the medical record confirming the DSM-V diagnosis of anxiety disorder including; separation anxiety disorder, generalized anxiety disorder, and/or social phobia. If this documentation is not present or is more than 2 years old, then the appropriate section of the K-SADS will be administered to confirm diagnosis.
3. At least moderate severity of anxiety symptoms as determined by score of ≥ 13 on the Pediatric Anxiety Rating Scale (PARS).
4. On a stable dose of psychotropic medications for at least one month, with no major changes projected.

Exclusion Criteria:

1. Presence of prominent diarrhea.
2. Diagnosis of diabetes mellitus.
3. Presence of active suicidal ideation and behavior or psychosis. B-SSRS ideation score greater than 1. B-SSRS behavior score greater than 0.
4. Weight less than 20 kg.
5. Known pregnancy.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
To measure the safety of myo-inositol, anxiety and mood symptoms will be measured using Clinical Global Impression Severity (CGI-S). | Weeks 1-12
  This assessment rates the clinician's view of the patient's anxiety severity prior to and after initiating myo-inositol. Scores range from 0-7. Higher scores mean worse outcome.
To measure the safety of myo-inositol, anxiety and mood symptoms will be measured using the Patient Global Index of Change Severity (PGIC-S). | Weeks 1-12
  This scale is a parent and child report tool that evaluates participants' anxiety and assesses if there has been a decline in clinical status. Answer options are "0-None", "1-Mild", "2-Moderate", and "3-Severe" and describe symptoms of anxiety. Higher scores mean worse outcome.
To measure the tolerability of myo-inositol, the number of participants who are able to remain on myo-inositol for the full treatment period (10-12 weeks) will be measured. | Weeks 1-14
  At study completion, the number of participants who remained on myo-inositol for the full 10-12 weeks will be counted.
To measure the tolerability of myo-inositol, the number of participants able to remain on the full dosage of myo-inositol for the full treatment period (10-12 weeks) will be measured. | Weeks 3-8
  Participants will be titrated up to the full dose of myo-inositol by Week 3 and will remain on the full dose for 6 weeks unless they cannot tolerate the dose. At study completion, the number of participants who remained on the full-dose of myo-inositol for the full 10-12 weeks will be counted.
To measure the safety and tolerability of myo-inositol, a change from baseline on the Physical Symptom Checklist (Side Effect Rating Scale) will be measured. | Weeks 1-14
  This assessment is a parent and child report measure. Its scores range from 0 to 60. Higher scores are indicative of more physical and psychological symptoms and worse outcome.
To measure the safety of myo-inositol, the Brief Suicide Severity Rating Scale (B-SSRS) will be measured at each visit. | Weeks 1-12
  The B-SSRS probes for suicidal thoughts and behavior. The scores for both categories range from 0-5. If participants score greater than 1 on B-SSRS ideation or greater than 0 on B-SSRS behavior, then they cannot be enrolled or remain in the study. Higher scores mean worse outcome.
To measure the safety of myo-inositol, a fingerstick blood test will be done to measure glucose levels at the first and final study visits. | Week 1 & Week 10-12
  A glucometer will be used to test the blood glucose levels of participants.
To measure the safety of myo-inositol, physical measurements (height and weight) will be obtained. | Weeks 1-12
  Myo-inositol is dosed by the weight of the participant. To make sure the participant is taking the correct dose, weight will be measured at each study visit. Height will only be measured at Week 1 to calculate BMI. Also, change in weight or BMI will be followed.

SECONDARY OUTCOMES:
To measure the effectiveness of myo-inositol for mood symptoms, a change from baseline on the Moods and Feelings Questionnaire (MFQ) will be evaluated. | Weeks 1-12
  The Mood and Feelings Questionnaire (MFQ) is a child and parent report questionnaire that measures depressive symptoms in children and young adults. Scores range from 0 to 66. Higher score are indicative of increased depressive symptom severity and worse outcome.
To measure the effectiveness of myo-inositol for anxiety symptoms, a change from baseline on Clinical Global Impression Improvement (CGI-I) will be evaluated. | Weeks 2-12
  This assessment rates the clinician's view of the patient's anxiety improvement after initiating myo-inositol. Scores range from 0-7. Higher scores mean worse anxiety symptoms.
To measure the effectiveness of myo-inositol for anxiety symptoms, a change from baseline on Clinical Global Impression Severity (CGI-S) will be evaluated. | Weeks 2-12
  This assessment rates the clinician's view of the patient's anxiety severity before and after initiating myo-inositol. Scores range from 0-7. Higher scores mean more anxiety symptoms.
To measure the effectiveness of myo-inositol for anxiety symptoms, a change from baseline on Brief Child Mania Rating Scale Parent Version (BCMRS-P) will be evaluated. | Week 1 & Weeks 10-12
  The BMRS-P is a 10-item inventory rated on a 4 point Likert type scale anchored by 0 (never/rare), 1 (sometimes), 2 (often), and 3 (very often). Its purpose is to measure changes in symptoms of pediatric bipolar disorder (PBD) as they change over time. Scores range from 0 to 30. Higher scores mean more symptom severity.
To measure the effectiveness of myo-inositol for anxiety symptoms, a change from baseline on the Patient Global Index of Change Improvement (PGIC-I) will be evaluated. | Weeks 2-12
  This scale evaluates participants' anxiety and assesses if there has been an improvement in clinical status. Answer options are "Much Improved", "Minimally Improved", "No Change", "Minimally Worse", and "Much Worse".
To measure the effectiveness of myo-inositol for anxiety symptoms, a change from baseline on the Patient Global Index of Change Severity (PGIC-S) will be evaluated. | Weeks 1-12
  This scale is a child and parent self-report instrument used to evaluate participants' anxiety and assesses if there has been a decline in clinical status. Answer options are "0-None", "1-Mild", "2-Moderate", and "3-Severe" and describe symptoms of anxiety. Higher scores mean more anxiety symptoms and worse outcome.
To measure the effectiveness of myo-inositol for anxiety symptoms, a change from baseline on the Self-Report for Childhood Related Emotional Disorders (SCARED) will be evaluated. | Weeks 1-12
  The SCARED is a child and parent self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder, and social phobia. The SCARED consists of 41 items and 5 factors that parallel the DSM-IV classification of anxiety disorders. Scores range from 0-82. Scores greater than or equal to 25 indicate the presence of an anxiety disorder and scores in different items indicate the type of anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Glick, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Child and Adolescent Bipolar Services-WPIC Bellefield, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request from other researchers, we will make available de-identified subject data, as appropriate.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared, as deemed appropriate, starting 6 months after completion of the study for a period of 5 years.
Access Criteria: Biomedical researcher involved in research activity in a related field and from an established research institution.

REFERENCES:
- [Background] Benjamin J, Agam G, Levine J, Bersudsky Y, Kofman O, Belmaker RH. Inositol treatment in psychiatry. Psychopharmacol Bull. 1995;31(1):167-75. PMID 7675981
- [Background] Benjamin J, Levine J, Fux M, Aviv A, Levy D, Belmaker RH. Double-blind, placebo-controlled, crossover trial of inositol treatment for panic disorder. Am J Psychiatry. 1995 Jul;152(7):1084-6. doi: 10.1176/ajp.152.7.1084. PMID 7793450
- [Background] Eden Evins A, Demopulos C, Yovel I, Culhane M, Ogutha J, Grandin LD, Nierenberg AA, Sachs GS. Inositol augmentation of lithium or valproate for bipolar depression. Bipolar Disord. 2006 Apr;8(2):168-74. doi: 10.1111/j.1399-5618.2006.00303.x. PMID 16542187
- [Background] Fux M, Levine J, Aviv A, Belmaker RH. Inositol treatment of obsessive-compulsive disorder. Am J Psychiatry. 1996 Sep;153(9):1219-21. doi: 10.1176/ajp.153.9.1219. PMID 8780431
- [Background] Levine J. Controlled trials of inositol in psychiatry. Eur Neuropsychopharmacol. 1997 May;7(2):147-55. doi: 10.1016/s0924-977x(97)00409-4. PMID 9169302
- [Background] Levine J, Barak Y, Gonzalves M, Szor H, Elizur A, Kofman O, Belmaker RH. Double-blind, controlled trial of inositol treatment of depression. Am J Psychiatry. 1995 May;152(5):792-4. doi: 10.1176/ajp.152.5.792. PMID 7726322
- [Background] Palatnik A, Frolov K, Fux M, Benjamin J. Double-blind, controlled, crossover trial of inositol versus fluvoxamine for the treatment of panic disorder. J Clin Psychopharmacol. 2001 Jun;21(3):335-9. doi: 10.1097/00004714-200106000-00014. PMID 11386498
- [Background] Silverstone PH, McGrath BM, Kim H. Bipolar disorder and myo-inositol: a review of the magnetic resonance spectroscopy findings. Bipolar Disord. 2005 Feb;7(1):1-10. doi: 10.1111/j.1399-5618.2004.00174.x. PMID 15654927